CLINICAL TRIAL: NCT02318771
Title: An Exploratory Study to Investigate the Immunomodulatory Activity of Radiation Therapy (RT) in Combination With MK-3475 in Patients With Recurrent/Metastatic Head and Neck, Renal Cell Cancer, Melanoma and Lung Cancer
Brief Title: Radiation Therapy and MK-3475 for Patients With Recurrent/Metastatic Head and Neck Cancer, Renal Cell Cancer, Melanoma, and Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14P.524; 2014-085 (Other: CCRRC); JT 6980 (Other: JeffTrial Number)
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Metastatic Renal Cell Cancer; Recurrent Head and Neck Carcinoma; Recurrent Lung Carcinoma; Recurrent Renal Cell Carcinoma; Recurrent Skin Carcinoma; Stage III Renal Cell Cancer; Stage IV Lung Cancer; Stage IV Skin Melanoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Lung Neoplasms; Melanoma | interventions — Radiotherapy; Radiation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A1: RT (1 fraction, 8 Gy) + MK-3475 (Experimental): Patients undergo RT on day 1 per standard of care and then undergo biopsy 3-10 days later. Beginning 0-7 days after biopsy, patients receive MK-3475 IV over 30 minutes on day 1. Courses of MK-3475 repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation Therapy (RT); Drug: MK-3475
- A2: RT (5 fractions, 4 Gy) + MK-3475 (Experimental): Patients undergo RT on days 1-5 and then undergo biopsy 3-10 days later. Beginning 0-7 days after biopsy, patients receive MK-3475 as in Arm A1.
  Interventions: Radiation: Radiation Therapy (RT); Drug: MK-3475
- B1: MK-3475 + RT (1 fraction, 8 Gy) + MK-3475 (Experimental): Patients receive one dose of MK-3475 IV over 30 minutes on day 1 and then undergo 1 fraction of RT. Patients then receive MK-3475 IV over 30 minutes in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Radiation Therapy (RT); Drug: MK-3475
- B2: MK-3475 + RT (5 fractions, 4 Gy) + MK-3475 (Experimental): Patients receive MK-3475 as in Arm B1 and undergo 5 fractions of RT.
  Interventions: Radiation: Radiation Therapy (RT); Drug: MK-3475

INTERVENTIONS:
Radiation: Radiation Therapy (RT) — Undergo RT
  Other Names: Radiation; Radiotherapy
Drug: MK-3475 — Given IV
  Other Names: Pembrolizumab; Keytruda; lambrolizumab

SUMMARY:
This randomized clinical trial studies radiation therapy and MK-3475 in treating patients with head and neck cancer, kidney cancer, melanoma, or lung cancer that has returned, has spread to other parts of the body, or cannot be removed by surgery. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as MK-3475, may block tumor growth by targeting certain cells and causing the immune system to attack the tumor. Studying the effects of MK-3475 with radiation therapy on the body may help doctors learn whether it may be an effective treatment for these solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the immunomodulatory activity of radiation therapy (RT) or RT in combination with anti-programmed cell death 1 (PD)-1 antibody (MK-3475) in patients with recurrent/metastatic head and neck cancer, renal cell cancer, melanoma and lung cancer.

SECONDARY OBJECTIVES:

I. To explore whether programmed cell death ligand 1 (PD-L1) expression is associated with treatment response to the combination of RT and PD-1 blockade in renal cell cancer (RCC), head and neck cancer (HNC), lung cancer and melanoma.

II. To explore whether circulating tumor cells can be used to determine PD-L1 expression.

III. To explore other immune-related biomarker changes after RT: soluble PD-L1, cytokines etc.

OUTLINE: Patients are randomized to 1 of 4 treatment arms.

ARM A1: Patients undergo radiation therapy on day 1 per standard of care and then undergo biopsy 3-10 days later. Beginning 0-7 days after biopsy, patients receive MK-3475 intravenously (IV) over 30 minutes on day 1. Courses of MK-3475 repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM A2: Patients undergo radiation therapy on days 1-5 and then undergo biopsy 3-10 days later. Beginning 0-7 days after biopsy, patients receive MK-3475 as in Arm A1.

ARM B1: Patients receive one dose of MK-3475 IV over 30 minutes on day 1 and then undergo 1 fraction of RT. Patients then receive MK-3475 IV over 30 minutes in the absence of disease progression or unacceptable toxicity.

ARM B2: Patients receive MK-3475 as in Arm B1 and undergo 5 fractions of RT.

After completion of study treatment, patients are followed up at approximately 30 days and then every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have provided tissue from an archival tissue sample ( < 6 months old) or newly obtained core biopsy of a tumor lesion before radiation therapy. A core biopsy will be required. It is mandatory to have post-radiation re-biopsy.
4. In addition to index lesion, there are ≥ 1 measurable lesion(s).
5. Have a performance status of ≤ 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function defined as the following:

   * Absolute neutrophil count (ANC) ≥1,500 /mcL
   * Platelets ≥100,000 / mcL
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
   * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.8 X upper limit of normal (ULN) OR

     ≥50 mL/min for subject with creatinine levels > 1.8 X institutional ULN
   * Serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
7. Female subjects of childbearing potential should have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 2 weeks of the radiation therapy.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the radiation therapy.
3. Has had a prior monoclonal antibody within 4 weeks prior to radiation therapy or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to radiation therapy or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Prior radiation therapy does not necessary excludes patients. The index lesion may be acceptable for stereotactic radiosurgery (SRS) and this will be determined by radiation oncologist.
   * Note: If there are more than one symptomatic lesions, patients will be excluded if the lesions can't be encompassed within one radiation portal.
   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer that has undergone potentially curative therapy.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the radiation therapy and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to radiation treatment.
7. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Has a known Human Immunodeficiency Virus infection (HIV 1/2 antibodies) or Acquired Immunodeficiency Syndrome((HIV/AIDS).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Has received a live vaccine within 30 days prior to the radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Change in PD-LI levels | Baseline to up to 10 days after last dose of RT
  Within each cohort, the significance of change in PD-L1 will be assessed using an exact one-sided sign test. The null hypothesis is that the average change (post-pre) is less than or equal to 0 while the alternative hypothesis is that the average change is greater than 0. The proportion of patients with improvement will be estimated along with an exact 95% confidence interval. As an exploratory analysis, the proportion will also be estimated separately within each cohort for the head and neck cancer patients.

SECONDARY OUTCOMES:
Response rate | Up to 4 years
  Summarized by treatment cohort along with exact 95% binomial confidence intervals.
Rate of toxicities | Up to 4 years
  Summarized by treatment cohort along with exact 95% binomial confidence intervals.
Progression-free survival | Up to 4 years
  Estimated by treatment cohort using the Kaplan-Meier method.
Biomarker levels | Up to 10 days after last dose of RT
  Repeated biomarker measurements will be modeled using mixed effects linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johnson, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Weber JS. Practical management of immune-related adverse events from immune checkpoint protein antibodies for the oncologist. Am Soc Clin Oncol Educ Book. 2012:174-7. doi: 10.14694/EdBook_AM.2012.32.79. PMID 24451730
- [Background] Weber JS, Kahler KC, Hauschild A. Management of immune-related adverse events and kinetics of response with ipilimumab. J Clin Oncol. 2012 Jul 20;30(21):2691-7. doi: 10.1200/JCO.2012.41.6750. Epub 2012 May 21. PMID 22614989
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Weber J, Thompson JA, Hamid O, Minor D, Amin A, Ron I, Ridolfi R, Assi H, Maraveyas A, Berman D, Siegel J, O'Day SJ. A randomized, double-blind, placebo-controlled, phase II study comparing the tolerability and efficacy of ipilimumab administered with or without prophylactic budesonide in patients with unresectable stage III or IV melanoma. Clin Cancer Res. 2009 Sep 1;15(17):5591-8. doi: 10.1158/1078-0432.CCR-09-1024. Epub 2009 Aug 11. PMID 19671877
- [Background] Lemech C, Arkenau HT. Novel treatments for metastatic cutaneous melanoma and the management of emergent toxicities. Clin Med Insights Oncol. 2012;6:53-66. doi: 10.4137/CMO.S5855. Epub 2012 Jan 5. PMID 22253555
- [Background] Phan GQ, Weber JS, Sondak VK. CTLA-4 blockade with monoclonal antibodies in patients with metastatic cancer: surgical issues. Ann Surg Oncol. 2008 Nov;15(11):3014-21. doi: 10.1245/s10434-008-0104-y. Epub 2008 Aug 21. PMID 18716842
- [Background] Bristol-Myers Squibb: YERVOY (ipilimumab): Serious and fatal immune- mediated adverse reactions-YERVOY Risk Evaluation and Mitigation Strategy (REMS). http://www.yervoy.com/hcp/rems.aspx
- [Background] Bristol-Myers Squibb: YERVOY (ipilimumab) prescribing information revised March 2011. http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/125377s0000lbl.pdf
- [Background] Janssen Biotech, Inc.: REMICADE (Infliximab) prescribing information revised September 2011. http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm?fuseaction=Search.La bel_Appr ovalHistory#labelinfo
- [Derived] Alexander GS, Palmer JD, Tuluc M, Lin J, Dicker AP, Bar-Ad V, Harshyne LA, Louie J, Shaw CM, Hooper DC, Lu B. Immune biomarkers of treatment failure for a patient on a phase I clinical trial of pembrolizumab plus radiotherapy. J Hematol Oncol. 2016 Sep 23;9(1):96. doi: 10.1186/s13045-016-0328-4. PMID 27663515
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/